CLINICAL TRIAL: NCT05277545
Title: The Effect of Technology Addiction Education Given to Nursing Students on Students' Perspectives and Addiction Levels
Brief Title: The Effect of Education on Technology Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KaratayUBK
Record Dates: First submitted 2022-01-28; First posted 2022-03-14 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-01

CONDITIONS: Technology Addiction
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect of teknology addiction training on the experimental group (Experimental): The arm explanations for which the analyzes of the research have not been completed yet cannot be made.
  Interventions: Behavioral: Technology addiction education
- Comparison of the experimental group and control group on technology addiction (Active Comparator): The arm explanations for which the analyzes of the research have not been completed yet cannot be made.
  Interventions: Behavioral: Technology addiction education

INTERVENTIONS:
Behavioral: Technology addiction education — Technology addiction personal development training was applied by the researcher to the students in the experimental group for 10 weeks.

SUMMARY:
The aim of this study is to determine the effect of the education given in technology addiction course to nursing students studying at a foundation university on students' perspectives on addiction and addiction levels.A self-report online survey method was used to collect data. After the data collection tools used were made suitable for filling in the online environment, the questionnaires were delivered to the participants using e-mail and social media networks. The pretest was collected just before the start of the personal development phase training on technology addiction. Then, technology addiction personal development training planned by the researcher was applied to the students in the experimental group for 10 weeks. After the end of the lessons, the same questionnaires were used as a posttest application. The same data collection tools were applied to the control group without any intervention.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of the education given in the technology addiction course to nursing students studying at a foundation university on the students' perspectives on addiction and addiction levels.Dependence; taking increasing amounts of a substance for purposes other than its intended purpose; It is the picture where the person cannot stop using even though it causes problems in his life and withdrawal symptoms appear when he reduces his substance intake. In addiction, the person continues to use the substance despite the problems related to family, social and work/school life (Koç, et al., 2018). Although not yet included in the DSM-5 diagnostic list, some conditions that are suggested to be candidates for inclusion in this list and that require further investigation have been identified. These conditions can be listed as "internet addiction", "social media addiction" and "smartphone addiction" (American Psychiatric Association, 2013.). Internet addiction constitutes the main framework of other internet-related addictions. In this context, it is emphasized that activities carried out on the Internet as well as the Internet are a source of addiction (Griffiths &, Szabo, 2014). Therefore, concepts such as "social media addiction", "digital game addiction" and "smartphone addiction" can be considered as addictions in which the active substance is the internet (Kwon, et al., 2013). Although a precise definition of the term "internet addiction", which was included in the DSM-5 for the first time, could not be made; It is defined as not being able to limit internet use, being stressed when internet access is blocked or restricted, spending time on the internet in increasing amounts, continuing to use the internet despite having problems in work/school life and family life. It is predicted that technological dependencies will take place more in the future versions of DSM (Savcı & Aysan, 2017).For this reason, it is inevitable to see the importance of intervening by determining students' perspectives on internet and technology addictions and their addiction levels, if any. At this point, the aim of the research is to see the effect of the education on technology addiction on students' perspectives and addiction levels.

hypotheses H1: Technology addiction education given to nursing students changes their perspectives on addiction.

H2: Technology addiction education given to nursing students positively affects their addiction assessments.

H3: Technology addiction education given to nursing students reduces the level of technology addiction.

Method:

Type of Study: This is a randomized controlled interventional study. Population and Sample of the Research The universe of this research will be all students studying in the nursing department at a foundation university in Konya. In the comparison of the experimental and control groups using the sample size power analysis of the research, the minimum number of subjects required in each group will be determined in order for the difference between them to be statistically significant in terms of scale scores. The experimental group of the research will consist of students who choose the elective technology addiction course, which has a chance of random selection. The control group will consist of students who have not chosen this course and have not taken a technology addiction course before.

Dependent and Independent Variables of the Research Dependent variables; students' perspectives on their own technology addiction and their level of technology addiction.

Independent variables; personal characteristics of students and technology addiction training to be given.Data Collection Method: An online survey method based on self-report will be used while collecting data. After these data collection tools to be used are made suitable for filling in the online environment, the questionnaires will be delivered to the participants using e-mail and social media networks. The pretest will be collected just before the start of the personal development training on technology addiction. After Dada, technology addiction personal development training planned by the researcher will be applied to the students in the experimental group for 10 weeks. After the end of the classes, the same questionnaires will be used as a posttest application.

Statistical Analysis of Data P<0.05 will be considered statistically significant by using the IBM SPSS Statistics 20.0 package program for the data obtained by statistical analysis from the questionnaires applied in the pretest and posttest phase of the research. In the association of demographic characteristics, the conformity of numerical values to the normal distribution will be checked. It is planned to use percentile, t-test in dependent groups, chi-square tests in nonparametric cases, Fisher Exact and Pearson chi-square tests in the analysis of the research.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student
* Studying in Nursing
* Volunteering to take the technology addiction course

Exclusion Criteria:

* Having a communication problem
* Receiving treatment for addiction
* Students undergoing psychiatric treatment

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Technology Addiction Scale | At the and of 5 month
  The scale to be used to evaluate this measure is the technology dependency scale. When interpreting the arithmetic averages of the whole scale, the 0-24 score range is "Not dependent", the 25-48 score range is "Low dependent", the 49-72 score range is "Moderately dependent", the 73-96 score range is "Highly Dependent", 97- The 120 point range is accepted as "Full Dependent". Cronbach Alpha values for the sub-dimensions of the scale were 0.786 for Social Network Addiction, 0.806 for Instant Messaging Addiction, 0.897 for Online Game Addiction, and 0.861 for Web Sites.Percentage, frequency and mean values will be used. To compare the results, the means obtained from the first and second measurements of the experimental and control groups will be compared with the t-test in the dependent groups.

SECONDARY OUTCOMES:
Personal Information Form | At the and of 5 month
  Personal information form prepared by using the literature; It consists of closed-ended questions with demographic characteristics. In the form created to evaluate the socio-demographic characteristics of the participants, there are questions about age, gender and students' perspectives on technology addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Dr Bayır, 1, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared with other researchers.

REFERENCES:
- [Derived] Bayir B, Topbas T. The effect of technology addiction training given to nursing students on the perspectives and addiction levels of students. Arch Psychiatr Nurs. 2023 Aug;45:152-157. doi: 10.1016/j.apnu.2023.06.012. Epub 2023 Jun 21. PMID 37544691